CLINICAL TRIAL: NCT05394974
Title: Evaluation of a Joint Consultation Between a Neurologist and a Clinical Psychologist, Dedicated to Neurodegenerative and/or Neurogenetic Disorders
Brief Title: Joint Consultation Between a Neurologist and a Clinical Psychologist
Acronym: JOCONDE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: JOCONDE
Record Dates: First submitted 2022-05-23; First posted 2022-05-27 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-05

CONDITIONS: Neurodegenerative Disorders
Keywords: Joint neurologist; psychologist consultation; neurodegenerative and/or neurogenetic disease
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Joint consultations appeared a few years ago in routine medical practice, but they are still not widely used and rarely evaluated.

The primary purpose of the study is to evaluate the impact for the patient of the presence of a clinical psychologist during the joint consultation.

The secondary purpose is to evaluate the impact for the patient and for the neurologist of the presence of a clinical psychologist during the joint consultation

ELIGIBILITY:
Inclusion Criteria:

* patient with a neurodegenerative and/or neurogenetic disease
* adult patient

Exclusion Criteria:

* dementia
* age <18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient with a neurodegenerative and/or neurogenetic disease
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction after the consultation assessed by 3 questions on a Likert scale | After consultation et 1 to 3 months later
  5-point Likert scale from which to select a response :
  1. Very satisfied.
  2. Moderately satisfied.
  3. Neither satisfied nor dissatisfied.
  4. Moderately dissatisfied.
  5. Very dissatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu ANHEIM, MD, PhD, Principal Investigator — Service de Neurologie - CHU de Strasbourg - France
Locations (1):
- Service de Neurologie - CHU de Strasbourg - France, Strasbourg, France